CLINICAL TRIAL: NCT05775783
Title: Effectiveness, Complications, and Mortality of Transvenous Lead Extraction in Patients With and Without Infections-Prospective Registry From a High-volume Center.
Brief Title: Effectiveness, Complications, and Mortality of TLE in Patients.
Acronym: EXTRACT
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Collaborators: Wojciech Wańha (Unknown)
Responsible Party: Principal Investigator, Kszysztof Gołba, Prof., Medical University of Silesia
Other Study IDs: 0001
Record Dates: First submitted 2023-02-25; First posted 2023-03-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Transvenous Lead Extraction
Keywords: Transvenous Lead Extraction; Cardiac Implantable Electronic Devices
MeSH Terms: interventions — Device Lead Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consecutive patients with CIEDs, treated with TLE (infections)
  Interventions: Procedure: Transvenous lead extraction
- Consecutive patients with CIEDs, treated with TLE (no-infections)
  Interventions: Procedure: Transvenous lead extraction

INTERVENTIONS:
Procedure: Transvenous lead extraction — Each TLE procedure was started using the single traction method. If this attempt was not sufficient to extract the lead, then the following methods were used: mechanical extraction sheaths (Byrd, Cook Vascular Inc., Leechburg, PA, USA), locking and nonlocking stylets (Liberator® Beacon® Tip Locking Stylet, Cook® Medical, Leechburg, PA, USA), powered extraction sheaths (Evolution or Evolution II Mechanical Dilator Sheath, Cook® Medical, Leechburg, PA, USA). A side retrieval snare loop (Needle's Eye Snare, Cook® Medical, Leechburg, PA, USA) was used for the femoral approach when the subclavian-only approach was insufficient.

SUMMARY:
The number of devices for cardiac pacing and defibrillation has increased in recent years. However, although they have improved in terms of quality and extended lifespan after implantation, they are not free from complications. The Achilles' heel of cardiac implantable electronic devices (CIEDs) is the risk of infections and lead failure, which, when untreated, can be the cause of poor outcomes and a high mortality rate. Abandoned leads predict serious adverse events, such as lead infections, death, electrical interference, or potential problems during future TLE procedures. Therefore, it is crucial to extract them, presuming the decision is warranted based on a patient's individual risk. TLE is a standard treatment for device-related complications, and while TLE procedures are relatively rare in comparison to the number of CIEDs that are implanted, the need for TLE has grown in recent years due to the aging population, an increasing number of upgrades of pacing systems, and a related rise in infection rates. According to the European Lead Extraction ConTRolled Registry (ELECTRa), the most frequent indication for TLE is CIED infection, with the majority of them being local infections. The second most common reason for TLE is lead dysfunction, which is observed in 38.1% of cases. In such cases, the treatment must be fast and effective. TLE is the first-line treatment for those patients and prevents further serious or even lethal complications. However, the goal of TLEis often to remove leads and also maintain access in the occluded vein by moving the sheath over the lead to the lead myocardial interface. TLE technology has recently shown substantial progress in improving the safety and effectiveness of the procedure. As a rule, single traction is the primary method of treatment, followed by more aggressive techniques such as locking stylet, mechanical sheaths, powered extraction sheaths, and femoral snares.

Data obtained in previous studies. indicated that identifying predictors of such undesirable adverse events appeared essential for optimizing the procedural technique. Another vital element to address were patients deemed at high risk of stricter follow-up and stronger secondary prevention strategies; notably, infected TLE patients have unique characteristics. The analysis of independent predictor outcomes could, thus, allow clinicians to better identify high-risk TLE patients. In light of this, the current registry aimed to investigate the composite short-term outcomes for infected and non-infected patients in real-world populations.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients who underwent TLE between 2016 and 2025 entered the EXTRACT Registry.

Exclusion Criteria:

- no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 702 patients
Sampling Method: Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Procedural success | 30 days
  Removing all targeted leads and their component parts without causing any permanently disabling complication or procedure-related death.
Clinical success | 30 days
  Removing all targeted leads and their component parts from the cardiovascular system or leaving a small part of the lead (<4cm) that did not adversely affect the objectives of the procedure or cause procedural-related death
Minor complications | 30 days
  Complications that did not require surgical intervention or involved minor surgical interventions that did not affect the patient's functionality.
All-cause death or occurrence of any major complication | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Krzysztof Gołba, Katowice, Poland

IPD SHARING:
Plan to Share IPD: Undecided